CLINICAL TRIAL: NCT06078540
Title: A Mobile Health (mHealth) Strategy for Improving Blood Pressure Control Among Adult Hypertensive African Americans
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB23-1110
Record Dates: First submitted 2023-10-05; First posted 2023-10-12 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Hypertension; Blood Pressure
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- USeeBP (Experimental): Participants will be asked to use the USeeBP mHealth app alongside participating in UCM-RPM program as part of their routine care.
  Interventions: Other: USeeBP

INTERVENTIONS:
Other: USeeBP — USeeBP is a low risk mobile medical app that proposes to do no more than:
  * Help patients (i.e., users) self-manage their disease or conditions without providing specific treatment or treatment suggestions;
  * Provide patients with simple tools to organize and track their health information;
  * Provide easy access to information related to patients' health conditions or treatments;
  * Help patients document, show, or communicate potential medical conditions to health care providers;

SUMMARY:
The purpose of this study is to test the proof-of-concept for adding a novel mHealth application, USeeBP, to the established UChicago Medicine Ambulatory Medicine Remote-Patient Monitoring (UCM-RPM) Hypertension Management Program in a population of African American adults with poorly controlled hypertension.

DETAILED DESCRIPTION:
This is a single-arm, proof of concept study, which we will use to assess for initial evidence of efficacy and technical feasibility of adding the USeeBP mHealth app as an adjunct to the UCM-RPM program.

This study integrates the USeeBP app into the existing UCM-RPM clinical pathway. Regular UCM-RPM program activities include monitoring home blood pressure (BP) measurement flowsheets, performing patient telephone and EPIC MyChart message outreach, and making medication adjustments. USeeBP is a secure, chat-based smartphone application. The app connects to a patient's electronic BP cuff (eCuff) via Bluetooth and sends BP data to the UCM-RPM program (rather than using the companion app to the eCuff that is used in the UCM-RPM program). The USeeBP app also allows the patient to set BP check and medication reminders, as well as provides patient education and opportunities to participate in healthy behavior challenges.

The primary study goal is to measure the effect of the USeeBP mobile app on home BP. Serial home blood pressure measurements will be collected at multiple time points. We hypothesize that there will be a decrease in BP across the study period.

ELIGIBILITY:
Inclusion Criteria:

* African American
* Ages 18 to 65 years old
* Able to demonstrate English reading literacy of at least 8th grade level [Rapid Estimate of Adult Literacy in Medicine, Revised (REALM-R) score ≥ 6]
* Prior hypertension (HTN) diagnosis
* Clinically measured SBP ≥ 160 mmHg recorded during at least 2 of last 4 encounters within past 2 years
* UCM-RPM Hypertension Management Program current or eligible participant
* Access to an Android or Apple iOS smartphone and its corresponding health app
* Access to an active data plan or home Wi-Fi
* Willing to use wireless electronic blood pressure cuff (eCuff)
* Has access to EPIC myChart mobile app or is willing to establish myChart account and download app
* Willing to download USeeBP study app to phone
* Willing to download and use USeeBP app with staff assistance

Exclusion Criteria:

* Hypertension is managed by a specialist (specialist prescribes the anti-hypertensive therapies)
* Baseline blood pressure greater than 180/110
* Prior enrollment in the study
* Known pregnancy
* Prisoners
* Active opioid dependency
* Homelessness
* Psychiatric hospitalization in the last year
* Serious existing medical conditions that may make BP control difficult or necessitate frequent hospitalization (cirrhosis or hepatic failure, stage IV or V chronic kidney disease, interstitial nephritis, pulmonary arterial hypertension, right heart failure, history of dementia or neurocognitive disability, advanced heart failure, organ transplant, immunosuppressive therapy, active cancer treatment, patients on hospice care), stroke or myocardial infarction in past 90 days, severe aortic stenosis
* Hospital admission for primary diagnosis of hypertensive emergency, hypertensive urgency, or uncontrolled hypertension in the past 90 days

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-10-27 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Change in home BP | Baseline, Week 12
  systolic pressure over diastolic pressure; measured by Bluetooth enabled, electronic, at home BP cuff

SECONDARY OUTCOMES:
Change in BP control rate | Baseline, Week 12
  measured by clinical BP cuff, BP control defined as clinically-measured BP < 140/90 mmHg
Change in medication adherence | Baseline, Week 12
  measured by Medication Adherence Report Scale (MARS-5); minimum value is 5, maximum value is 25; lower values indicate worse medication adherence
Number of EPIC myChart patient-provider messages and replies | Week 12
  total number of messages and replies
Number of hypertension related unscheduled emergency department or urgent care visits | Week 12
  total number of visits

CONTACTS AND LOCATIONS:
Overall Officials: David G. Beiser, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States